CLINICAL TRIAL: NCT00378209
Title: Am Open-Label Phase II Study of the Safety and Efficacy of Bortezomib, Lenalidomide, and Dexamethasone Combination Therapy for Patients With Relapsed or Relapsed and Refractory Multiple Myeloma
Brief Title: Bortezomib, Lenalidomide, and Dexamethasone Combination Therapy for Patients With Relapsed or Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Celgene Corporation (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Paul G. Richardson, MD, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-147
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Myeloma
Keywords: relapsed multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Dexamethasone

ARMS (1):
- lenalidomide, dexamethasone, bortezomib combination (Experimental): Participants took the study medication in the clinic on Cycle 1 day 1. Each treatment cycle lasted three weeks. They took the lenalidomide (capsules) every day for the first two weeks only (days 1-14). They took the dexamethasone (tablets) on Day 1, 2, 4, 5, 8, 9, 11 and 12 and came to the outpatient treatment center for intravenous bortezomib on Day 1, 4, 8 and 11. The third week of the cycle was a rest period and the participant did not take any study medication.
  Interventions: Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Given intravenously on days 1,4,8 and 11 of a 21-day cycle for a minimum of 8 cycles.
Drug: Lenalidomide — Taken orally once a day for 2 weeks (days 1-14) of a 21-day cycle for a minimum of 8 cycles
Drug: Dexamethasone — Taken orally on days 1,2,4,5,8,9,11,and 12 of a 21-day cycle for a minimum of 8 cycles

SUMMARY:
The purpose of this study is to evaluate the effectiveness and side effects of the bortezomib, lenalidomide and dexamethasone combination in relapsed or relapsed and refractory multiple myeloma. Each of these drugs are approved by the U.S Food and Drug Administration, but have not been approved in the combination for treating patients in this setting.

DETAILED DESCRIPTION:
* Participants took the study medication in the clinic on Cycle 1 day 1. Each treatment cycle lasted three weeks. They took the lenalidomide (capsules) every day for the first two weeks only (days 1-14). They took dexamethasone (tablets) on Day 1, 2, 4, 5, 8, 9, 11 and 12 and came to the outpatient treatment center for intravenous bortezomib on Day 1, 4, 8 and 11. The third week of the cycle was a rest period and the participant did not take any study medication.
* Certain tests and procedures were performed throughout each treatment cycle at definitive time periods. These tests included: medical history update, physical/neurological examination, skeletal survey (x-rays or scan), blood samples, urine samples, optional bone marrow aspiration/tissue biopsy, 12-lead ECG, and MRI/CT (if needed).
* It was expected that participants were going to complete at least 8 cycles of the study, which adds up to 168 days. If the participant completed the first 8 cycles, had stable or responding disease and had not experienced bad side effects, they were allowed to continue treatment on a maintenance schedule, detailed in the protocol, at the study doctor's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma based on standard diagnostic criteria or by the new International Myeloma Foundation 2003 Diagnostic Criteria
* Relapsed or relapsed and refractory disease after receiving between 1 and 3 prior regimens
* Negative serum or urine pregnancy test
* Age 18 years or older
* Karnofsky performance status of 60 or greater

Exclusion Criteria:

* Grade 2 or greater peripheral neuropathy within 14 days before enrollment
* Renal insufficiency (serum creatinine > 2.5 mg/dL)
* Evidence of mucosal or internal bleeding and/or platelet refractory
* ANC < 1000 cells/mm3
* Hemoglobin < 8.0 g/dL
* AST or ALT greater than or equal to 2 x ULN
* Concomitant therapy medications that include corticosteroids
* Myocardial infarction within 6 months prior to enrollment or has NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Clinically relevant active infection or serious co-morbid medical conditions
* Prior malignancy (within last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or breast cancer, in situ prostate cancer
* Pregnant or breast-feeding
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Uncontrolled diabetes mellitus
* Hypersensitivity to acyclovir or similar anti-viral drug
* POEMS syndrome
* Known HIV infection
* Known active hepatitis B or C viral infection
* Known intolerance to steroid therapy
* Subjects with primary refractory disease, defined as progression during initial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-08; Primary Completion 2012-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Richardson PG, Xie W, Jagannath S, Jakubowiak A, Lonial S, Raje NS, Alsina M, Ghobrial IM, Schlossman RL, Munshi NC, Mazumder A, Vesole DH, Kaufman JL, Colson K, McKenney M, Lunde LE, Feather J, Maglio ME, Warren D, Francis D, Hideshima T, Knight R, Esseltine DL, Mitsiades CS, Weller E, Anderson KC. A phase 2 trial of lenalidomide, bortezomib, and dexamethasone in patients with relapsed and relapsed/refractory myeloma. Blood. 2014 Mar 6;123(10):1461-9. doi: 10.1182/blood-2013-07-517276. Epub 2014 Jan 15. PMID 24429336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 65 eligible participants were enrolled from the 6 institutions in the United States between September 2006 and April 2008 and 64 out of 65 received protocol treatment.
Pre-assignment Details: Participants screened over a 3 week period.
Groups:
- Lenalidomide, Dexamethasone, Bortezomib Combination: Patients were treated for up to 8 21-day cycles with the combination of bortezomib 1.0 mg/m2 IV, days 1, 4, 8, and 11, and oral lenalidomide 15 mg/day, days 1 through 14, with oral dexamethasone 40 mg/day (cycles 1-4) and 20 mg/day (cycles 5-8) on the days of and days after bortezomib dosing (days 1, 2, 4, 5, 8, 9, 11, and 12).Following a protocol amendment , dexamethasone dosing was reduced to 20 mg/day in cycles 1 through 4 and 10 mg/day in cycles 5 through 8.
  Beyond cycle 8, responding patients and those with stable disease (SD) could receive maintenance therapy until disease progression or unacceptable toxicity. Maintenance therapy comprised bortezomib and lenalidomide at the doses tolerated on completion of cycle 8, with lenalidomide on days 1 through 14 and using an amended schedule of weekly bortezomib (days 1 and 8) and dexamethasone 10 mg on days 1, 2, 8, and 9.
Period: Overall Study
Arm/Group | Lenalidomide, Dexamethasone, Bortezomib Combination
Started | 64 (1 patient who never started treatment was excluded in the analysis.)
Completed | 42 (This included patients who completed at least 8 cycles of combination therapy with all drugs.)
Not Completed | 22
Not completed — Progressive disease | 11
Not completed — Adverse Event | 3
Not completed — Initiation of non-protocol therapy | 3
Not completed — Physician Decision | 3
Not completed — Death | 1
Not completed — Treatment delay | 1

BASELINE CHARACTERISTICS:
Population: 65 patients were enrolled and 64 were treated. One patient who was never treated was excluded from the analysis.
Arm/Group | Lenalidomide, Dexamethasone, Bortezomib Combination
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 65 [32 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Alive and Without Progressive Disease (PD) for ≥6 Months
Description: Response assessed by the European Group for Blood and Marrow Transplant (EBMT) criteria, modified to include nCR and VGPR from the international uniform response criteria (IMWG).
  Progressive disease (PD) required one or more of the following:
  >25% increased in serum monoclonal paraprotein (must also be an absolute increase of at least 5 g/L and confirmed on a repeat investigation) >25% increased in 24-hour urinary light chain excretion (must also be an absolute increase of at least 200 mg/24 h and confirmed on a repeat investigation) >25% increased in plasma cells in a bone marrow aspirate or on trephine biopsy (must also be an absolute increase of at least 10%) Definite increase in the size of existing lytic bone lesions or soft tissue plasmacytomas.
  Development of new bone lesions or soft tissue plasmacytomas (not including compression fracture).
  Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.8 mmol/L not attributable to any other cause).
Time Frame: 6 months after therapy
Measure: Number (90% Confidence Interval); unit: percentage of treated patients
Arm/Group | Lenalidomide, Dexamethasone, Bortezomib Combination
Number analyzed (Participants) | 64
percentage of treated patients | 75 [65 to 84]

2. Secondary Outcome: Objective Response Rate
Description: Response assessed by the European Group for Blood and Marrow Transplant (EBMT) criteria, modified to include nCR and VGPR from the international uniform response criteria (IMWG).
  Objective response was defined by the achievement of at least Partial Response (PR) or better (CR-complete response, nCR-near complete response, and VGPR-very good partial response).
Time Frame: Assessed every cycle for up to 8 cycles and best response was reported
Measure: Number (90% Confidence Interval); unit: percentage of treated patients
Arm/Group | Lenalidomide, Dexamethasone, Bortezomib Combination
Number analyzed (Participants) | 64
percentage of treated patients | 64 [53 to 74]

3. Secondary Outcome: Duration of Response
Description: Duration of response will be measured as the time from initiation of a response to first documentation of disease progression or death, or date last known progression-free and alive for those who have not progressed or died.
Time Frame: Assessed at a median follow-up of 44 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide, Dexamethasone, Bortezomib Combination
Number analyzed (Participants) | 64
months | 8.7 [6.6 to 11.1]

4. Secondary Outcome: Progression Free Survival
Description: Progression-free survival is defined as the time from registration to the disease progression or death from any cause, censored at date last known progression-free for those who have not progressed or died.
Time Frame: aassesed at a median follow-up of 44 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide, Dexamethasone, Bortezomib Combination
Number analyzed (Participants) | 64
months | 9.5 [7.2 to 11.7]

5. Secondary Outcome: Overall Survival
Description: defined as time from treatment initiation to death, or last known to be alive for those who had not died
Time Frame: assesed at a median follow-up of 44 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Lenalidomide, Dexamethasone, Bortezomib Combination
Number analyzed (Participants) | 64
month | 30 [24 to 37]

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment (including both 8 cycles of combination therapy and maintenance therapy) and for 30 days after the end of treatment
Arm/Group | Lenalidomide, Dexamethasone, Bortezomib Combination
Serious Adverse Events (participants affected / at risk) | 47/64
Other Adverse Events (participants affected / at risk) | 34/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide, Dexamethasone, Bortezomib Combination (N=64)
Fatigue (General disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 19
Diarrhea (Gastrointestinal disorders) | 2 — w/o prior colostomy
hyperglycemia (Metabolism and nutrition disorders) | 6
peripheral edema (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Pain: extremity (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 6
Motor Neuropathy (Nervous system disorders) | 2
rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Dizziness (General disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 5
Pulmonary/ Upper Respiratory Event (Respiratory, thoracic and mediastinal disorders) | 4
Atrial Fibrillation (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 1
Lung Infection (Infections and infestations) | 1 — With concurrent grade 0-2 Neutropenia
Confusion (Psychiatric disorders) | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Psychosis (Psychiatric disorders) | 1
Fever (General disorders) | 1 — Without Neutropenia
Hypophosphatemia (Metabolism and nutrition disorders) | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide, Dexamethasone, Bortezomib Combination (N=64)
Sensory Neuropathy (Nervous system disorders) | 34
Fatigue (General disorders) | 29
Neutropenia (Blood and lymphatic system disorders) | 8
Diarrhea (Gastrointestinal disorders) | 24 — Without prior colostomy
Muscle Pain (Musculoskeletal and connective tissue disorders) | 25
Hyperglycemia (Metabolism and nutrition disorders) | 18
Peripheral Edema (Blood and lymphatic system disorders) | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Constipation (Gastrointestinal disorders) | 19
Insomnia (General disorders) | 18
Extremity Pain (General disorders) | 14
Anemia (Blood and lymphatic system disorders) | 14
Nausea (Gastrointestinal disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 5
Neuropathic Pain (Nervous system disorders) | 11
Rash/ desquamation (Skin and subcutaneous tissue disorders) | 8
Dizziness (General disorders) | 8
Fever (General disorders) | 6 — without concurrent neutropenia
Motor Neuropathy (Nervous system disorders) | 7
Infection (Infections and infestations) | 15
Anorexia (Endocrine disorders) | 8
agitation (Nervous system disorders) | 8
depression (Nervous system disorders) | 7
hypokalemia (Endocrine disorders) | 7
neurologic- other (Nervous system disorders) | 7
hypoglycemia (Metabolism and nutrition disorders) | 6
joint pain (Musculoskeletal and connective tissue disorders) | 6
anxiety (Nervous system disorders) | 5
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
hypomagnesemia (Metabolism and nutrition disorders) | 5
Blurred vision (Eye disorders) | 5
vomiting (Gastrointestinal disorders) | 5
aspartate transaminase disorder (Metabolism and nutrition disorders) | 4
dyspepsia (Gastrointestinal disorders) | 4
nonneuropatic generalized weakness (Musculoskeletal and connective tissue disorders) | 4
weight gain (Metabolism and nutrition disorders) | 4
alanine aminotransferase disorder (Metabolism and nutrition disorders) | 3
abdominal pain (Gastrointestinal disorders) | 3
alkaline phosphatase disorder (Metabolism and nutrition disorders) | 3
cough (Respiratory, thoracic and mediastinal disorders) | 3
cushingnoid appearance (Endocrine disorders) | 3
ocular- other (Eye disorders) | 3
tinnitus (Ear and labyrinth disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days